CLINICAL TRIAL: NCT01249053
Title: Expression of Optic Atrophy Type 1 (OPA1) Protein in Lung Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Fang Hsin-Yuan/Director, China Medical University Hospital
Other Study IDs: DMR99-IRB-062
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-11

CONDITIONS: Lung Adenocarcinoma
Keywords: OPA1; lung adenocarcinomas; Prognosis; Expression of optic atrophy type 1 (OPA1) protein in lung adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Optic atrophy type 1(OPA1) is a nuclear dynamin-related GTPase, targeted to the inner mitochondrial membrane, which plays a role in mitochondrial fusion. Mitochondria fusion is associated with process of apoptosis. . OPA1 plays an important role in the mitochondrial bioenergetics and mitochondrial networks. The changes in mitochondrial shape and mitochondrial bioenergetics may be cause of the disease. In this study, we investigate the expression of OPA1 in lung adenocarcinoma (LADC) cells and tissue.

ELIGIBILITY:
Inclusion Criteria:

* We will collect paraffin blocked resected lung tissue samples from stage I~IIIa non-small cell lung cancer patients (age, 40~80 years old) who received lobectomy of the affected lung.

Exclusion Criteria:

* History of uremia, other malignant disease, and liver cirrhosis
* History of pneumonia and pulmonary tuberculosis
* History of long period of medications.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 2006 and December 2008, we will retrospectively enroll 100 consecutive LADC patients who were admitted to the Department of Thoracic Surgery of China Medical University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-08

CONTACTS AND LOCATIONS:
Locations (1):
- Fang Hsin Yuan, Taichung, Taiwan